CLINICAL TRIAL: NCT03334734
Title: Multicenter, Open, Randomized Study With Active Control to Evaluate the Early Bactericidal Activity, Safety and Pharmacokinetics of the Drug PBTZ169 When Used in Patients With First-diagnosed Tuberculosis of the Respiratory System With Bacterial Excretion and Saved Bacterial Susceptibility to Isoniazid and Rifampicin
Brief Title: Phase 2a Study of PBTZ169
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Very slow enrollment
Sponsor: Nearmedic Plus LLC (Industry)
Collaborators: OCT LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PBTZ169-A15-C2A-1
Record Dates: First submitted 2017-11-03; First posted 2017-11-07 (Actual); Results first posted 2020-03-09 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-02

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; PBTZ169; antimycobacterial
MeSH Terms: conditions — Tuberculosis | interventions — macozinone; Isoniazid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PBTZ169, 160 mg (Experimental): 2 capsules 80 mg of PBTZ169 once a day for 14 days
  Interventions: Drug: PBTZ169
- PBTZ169, 320 mg (Experimental): 4 capsules 80 mg of PBTZ169 once a day for 14 days
  Interventions: Drug: PBTZ169
- PBTZ169, 640 mg (Experimental): 8 capsules 80 mg of PBTZ169 once a day for 14 days
  Interventions: Drug: PBTZ169
- Isoniazid, 600 mg (Active Comparator): 2 tablets 300 mg of Isoniazid once a day for 14 days
  Interventions: Drug: Isoniazid

INTERVENTIONS:
Drug: PBTZ169 — Once a day for 14 days
  Arms: PBTZ169, 160 mg; PBTZ169, 320 mg; PBTZ169, 640 mg
Drug: Isoniazid — Once a day for 14 days
  Arms: Isoniazid, 600 mg

SUMMARY:
Multicenter, open, randomized study with active control (isoniazid) to evaluate the early antibacterial activity, safety and pharmacokinetics of the drug PBTZ169 (capsules 80 mg) when used in patients with first-diagnosed tuberculosis of the respiratory system with bacterial excretion and saved bacterial susceptibility to isoniazid and rifampicin

DETAILED DESCRIPTION:
This phase 2a study is aimed to evaluate the early bactericidal activity of a new anti-tuberculosis drug PBTZ169 (capsules 80 mg), and its results will allow preliminary evaluate antimycobacterial properties of PBTZ169 and confirm a potentially more effective dose for subsequent studies. This study is an open, randomized comparative efficacy (on the parameter of early bactericidal activity), safety and pharmacokinetics study of PBTZ169 in patients with first-diagnosed lung tuberculosis and preserved sensitivity to base antimycobacterial drugs: rifampicin and isoniazid.

Within the framework of the study, it is planned to use the studied drugs (PBTZ169 and isoniazid) as monotherapy within 14 days. Isoniazid is used as a "positive control", that is, in order to determine whether the method of assessing efficacy on the parameter of early bactericidal activity is working.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent received from a volunteer
* Men and women aged 18 to 65 years, inclusive
* The first-diagnosed active pulmonary tuberculosis, confirmed by characteristic radiographic changes (infiltration, dissemination, destruction) during radiography or computed tomography of chest organs, without damage to other organs or with the defeat of one or more of the following organs: larynx, trachea, bronchi, lymph nodes
* The amount of sputum given by the patient is sufficient for carrying out the analyzes provided for by the protocol, but not less than 4-5 ml at the screening
* The presence of acid-fast mycobacteria in the sputum according to the results of microscopy of smears (1+ and more using the method of microscopy with luminescent dye staining according to the Order of the Ministry of Health of the Russian Federation of March 21, 2003 No. 109, the last edition) and the detection of the DNA of mycobacteria of tuberculosis by the results of molecular genetic methods of diagnosis
* Body weight not less than 51 kg
* Body mass index of 18.5-25 kg/m2
* Ability, according to investigators opinion, to comply with all requirements of the protocol
* Agreement to use double contraception method during the study participation and for 3 months after the test drug administration - combination of male condom with not less than one of the following methods:

  * female partner using hormonal contraception;
  * using aerosols, creams, suppositories and other agents containing spermicides;
  * female partner using intrauterine device

Exclusion Criteria:

* Extrapulmonary localization of tuberculosis
* Presence of resistance to rifampicin and / or isoniazid in the study of sputum samples using molecular genetic methods
* Admission of any anti-tuberculosis drugs from the moment of diagnosis of tuberculosis to the moment of inclusion in the study
* The presence of absolute indications for surgical treatment of tuberculosis at the time of screening
* Positive tests for serological markers of syphilis or HIV infection during screening; active hepatitis or decompensated hepatic cirrhosis
* Aggravated allergic history, including presence of at least one episode of drug allergy
* The values of renal and / or hepatic parameters according to laboratory analyzes (taking into account the range of normal laboratory values):

  * Aspartate aminotransferase (AST) level > 2.0 x upper limit of the norm
  * Alanine aminotransferase (ALT) level > 2.0 x upper limit of norm
  * General bilirubin level > 1.5 x upper limit of norm
  * Creatinine level > 1.5 x upper limit of norm
* Individual drug components intolerance
* Presence in the anamnesis of malignant neoplasms, except for basal cell skin cancer
* The presence of severe chronic somatic diseases in the stage of decompensation, including diseases of the cardiovascular, bronchopulmonary, neuroendocrine system, ear, nose and throat (ENT) organs, the gastrointestinal tract, liver, kidneys, blood, skin, or any other somatic or mental diseases that, according to the researcher, prevent the patient from entering the study
* Gastrointestinal surgeries (except for appendectomy performed not less than 1 year before screening)
* Mental illness that may interfere with the patient's compliance with the protocol
* Diabetes mellitus
* Acute viral and bacterial infections at the time of enrollment or within 2 weeks before enrollment
* Alcoholism (except in cases when the patient is able, in the opinion of the researcher, to refrain from taking alcohol during the period of participation in the study), drug addiction, abuse of medicines
* Positive tests for narcotic and psychotropic agents
* Regular admission or use (including externally) of any hormonal medicines lasting more than 1 week less than 30 days before screening (with the exception of oral hormonal contraceptives and intrauterine spirals containing hormones)
* Use of cytostatic drugs less than 30 days before screening
* Multiple admission of drugs with the described in the instructions for medical use adverse events related to nervous system, hemodynamic and hepatic functions with frequencies "very frequent" (≥10%) and "often" (≥1% and <10%) less than 21 days before screening
* Pregnancy or lactation period
* Planned conception or sperm donation during the study after the test drug administration or during 3 months after the last date of drug administration
* Participation in other clinical studies of drugs within less than 3 months before the screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-12-16 (Actual); Primary Completion 2017-09-10 (Actual); Study Completion 2018-02-22 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PBTZ169, 160 mg | PBTZ169, 320 mg | PBTZ169, 640 mg | Isoniazid, 600 mg
Started | 4 | 4 | 7 | 1
Completed | 4 | 4 | 5 | 1
Not Completed | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PBTZ169, 160 mg | PBTZ169, 320 mg | PBTZ169, 640 mg | Isoniazid, 600 mg | Total
Number analyzed (Participants) | 4 | 4 | 7 | 1 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.0 (13.0) | 48.8 (10.7) | 43.7 (14.8) | 41.0 (0) | 46.1 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 2 | 0 | 2
  Male | 4 | 4 | 5 | 1 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 4 | 4 | 7 | 1 | 16
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Russia | 4 | 4 | 7 | 1 | 16

OUTCOME MEASURES:

1. Primary Outcome: Early Bactericidal Activity (0-14)
Description: Early bactericidal activity 14 days from the monotherapy start date (EBA 0-14): agar inoculation, the mean of two measurements at the Visit
Time Frame: 14 days after the onset of monotherapy
Population: FAS
Measure: Mean (Standard Deviation); unit: CFU per 1 mL of sputum
Arm/Group | PBTZ169, 160 mg | PBTZ169, 320 mg | PBTZ169, 640 mg | Isoniazid, 600 mg
Number analyzed (Participants) | 4 | 4 | 7 | 1
CFU per 1 mL of sputum | 0.061 (0.085) | 0.015 (0.025) | 0.071 (0.126) | 0.237 (0)

2. Primary Outcome: Early Bactericidal Activity (0-14)
Description: Early bactericidal activity 14 days from the monotherapy start date (EBA 0-14): PCR, the mean of two measurements at the Visit
Time Frame: 14 days after the onset of monotherapy
Population: FAS
Measure: Mean (Standard Deviation); unit: cell count per 1 mL of sputum
Arm/Group | PBTZ169, 160 mg | PBTZ169, 320 mg | PBTZ169, 640 mg | Isoniazid, 600 mg
Number analyzed (Participants) | 4 | 4 | 7 | 1
cell count per 1 mL of sputum | 0.038 (0.081) | -0.014 (0.048) | 0.097 (0.136) | -0.099 (0)

3. Secondary Outcome: Early Bactericidal Activity (0-2)
Description: EBA (0-2): agar inoculation, the mean of two measurements at the Visit
Time Frame: 2 days after the onset of monotherapy
Population: FAS
Measure: Mean (Standard Deviation); unit: CFU per 1 mL of sputum
Arm/Group | PBTZ169, 160 mg | PBTZ169, 320 mg | PBTZ169, 640 mg | Isoniazid, 600 mg
Number analyzed (Participants) | 4 | 4 | 7 | 1
CFU per 1 mL of sputum | 0.496 (0.615) | 0.124 (0.095) | -0.003 (0.452) | -0.243 (0)

4. Secondary Outcome: Early Bactericidal Activity (0-7)
Description: EBA (0-7): agar inoculation, the mean of two measurements at the Visit
Time Frame: 7 days after the onset of monotherapy
Population: FAS
Measure: Mean (Standard Deviation); unit: CFU per 1 mL of sputum
Arm/Group | PBTZ169, 160 mg | PBTZ169, 320 mg | PBTZ169, 640 mg | Isoniazid, 600 mg
Number analyzed (Participants) | 4 | 4 | 7 | 1
CFU per 1 mL of sputum | 0.078 (0.136) | 0.026 (0.069) | 0.064 (0.102) | 0.090 (0)

5. Secondary Outcome: Early Bactericidal Activity (0-2)
Description: EBA (0-2): PCR, the mean of two measurements at the Visit
Time Frame: 2 days after the onset of monotherapy
Population: FAS
Measure: Mean (Standard Deviation); unit: cell count per 1 mL of sputum
Arm/Group | PBTZ169, 160 mg | PBTZ169, 320 mg | PBTZ169, 640 mg | Isoniazid, 600 mg
Number analyzed (Participants) | 4 | 4 | 7 | 1
cell count per 1 mL of sputum | -0.110 (0.872) | 0.007 (0.084) | 0.085 (0.397) | 0.627 (0)

6. Secondary Outcome: Early Bactericidal Activity (0-7)
Description: EBA (0-7): PCR, the mean of two measurements at the Visit
Time Frame: 7 days after the onset of monotherapy
Population: FAS
Measure: Mean (Standard Deviation); unit: cell count per 1 mL of sputum
Arm/Group | PBTZ169, 160 mg | PBTZ169, 320 mg | PBTZ169, 640 mg | Isoniazid, 600 mg
Number analyzed (Participants) | 4 | 4 | 7 | 1
cell count per 1 mL of sputum | -0.044 (0.076) | -0.004 (0.081) | 0.116 (0.186) | -0.408 (0)

7. Secondary Outcome: Peak Plasma Concentration (Сmax) of PBTZ169
Description: Peak plasma concentration (Сmax) of PBTZ169 for multiple dosing
Time Frame: Up to 72 hours after the last drug administration
Population: PKA: the pharmacokinetic analysis population for multiple dosing comprised all patients participating in the PK study who had received at least one dose of the study drug PBTZ169, provided that data on study drug concentration (with at least one measurement above BLQ) was available.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | PBTZ169, 160 mg | PBTZ169, 320 mg | PBTZ169, 640 mg
Number analyzed (Participants) | 4 | 4 | 7
ng/ml | 34.4714 (18.6498) | 122.0135 (96.3347) | 101.3818 (31.3830)

8. Secondary Outcome: Minimal Plasma Concentration (Сmin) of PBTZ169
Description: Minimal plasma concentration (Сmin) of PBTZ169: concentration measurement following single dosing
Time Frame: for single dosing , Day 1 (24 h after 1st dose of PBTZ169)
Population: PKA
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | PBTZ169, 160 mg | PBTZ169, 320 mg | PBTZ169, 640 mg
Number analyzed (Participants) | 4 | 4 | 7
ng/ml | 0.4985 (0.4475) | 0.2678 (0.3375) | 1.0275 (0.9101)

9. Secondary Outcome: Residual Concentration (Ctrough) of PBTZ169
Description: Residual concentration (Ctrough) of PBTZ169, measured 24 hours after the first dose administration, prior to the last dose, and 24 hours after the last dose
Time Frame: Up to 72 hours after the last drug administration
Population: PKA
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | PBTZ169, 160 mg | PBTZ169, 320 mg | PBTZ169, 640 mg
Number analyzed (Participants) | 4 | 4 | 7
ng/ml
  24 hours after the first dose (Ctrough_SD24) | 0.7835 (0.6820) | 1.4116 (1.2712) | 1.8712 (0.9453)
  prior to the last dose (Ctrough_MD0) | 2.1610 (1.6332) | 4.9505 (1.4050) | 18.2674 (27.2441)
  24 hours after the last dose (Ctrough_MD24) | 1.4207 (1.0145) | 2.9274 (1.4535) | 5.2710 (2.5201)

10. Secondary Outcome: Minimal Plasma Concentration (Сmin) of PBTZ169
Description: Minimal plasma concentration (Сmin) of PBTZ169: multiple dosing
Time Frame: Up to 72 hours after the last drug administration
Population: PKA
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | PBTZ169, 160 mg | PBTZ169, 320 mg | PBTZ169, 640 mg
Number analyzed (Participants) | 4 | 4 | 5
ng/ml | 1.4207 (1.0145) | 3.3889 (2.0001) | 4.9322 (2.4003)

11. Secondary Outcome: Time to Reach Maximum Concentration (Tmax) of PBTZ169
Description: Time to reach maximum concentration (Tmax) of PBTZ169 after single oral administration in different doses
Time Frame: for single dosing , Day 1 (24 h after 1st dose of PBTZ169)
Population: PKA
Measure: Median (Full Range); unit: h
Arm/Group | PBTZ169, 160 mg | PBTZ169, 320 mg | PBTZ169, 640 mg
Number analyzed (Participants) | 4 | 4 | 7
h | 1.250 [0.67 to 2.00] | 2.250 [1.00 to 6.00] | 2.000 [0.33 to 3.00]

12. Secondary Outcome: Time to Reach Maximum Concentration (Tmax) of PBTZ169
Description: Time to reach maximum concentration (Tmax) of PBTZ169 after multiple oral administration in different doses
Time Frame: Up to 72 hours after the last drug administration
Population: PKA
Measure: Median (Full Range); unit: h
Arm/Group | PBTZ169, 160 mg | PBTZ169, 320 mg | PBTZ169, 640 mg
Number analyzed (Participants) | 4 | 4 | 5
h | 2.000 [0.67 to 2.98] | 2.000 [1.00 to 6.00] | 1.500 [0.00 to 2.4]

13. Secondary Outcome: AUC(0-24)
Description: Area under the plasma concentration of PBTZ169 versus time curve in frames [0-24 hours]
Time Frame: Up to 24 hours after the first drug administration
Population: PKA
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | PBTZ169, 160 mg | PBTZ169, 320 mg | PBTZ169, 640 mg
Number analyzed (Participants) | 4 | 4 | 7
ng*h/ml | 93.604 (74.3008) | 120.954 (44.7920) | 237.153 (111.4025)

14. Secondary Outcome: Peak Plasma Concentration (Сmax) of PBTZ169
Description: Peak plasma concentration (Сmax) of PBTZ169: concentration measurement following single dosing
Time Frame: for single dosing , Day 1 (24 h after 1st dose of PBTZ169)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | PBTZ169, 160 mg | PBTZ169, 320 mg | PBTZ169, 640 mg
Number analyzed (Participants) | 4 | 4 | 7
ng/ml | 24.6543 (18.8506) | 35.5370 (23.4983) | 79.6684 (49.1865)

15. Secondary Outcome: AUC(0-24)
Description: Area under the plasma concentration of PBTZ169 versus time curve in frames [0-24 hours] for the last dosing (Day 14)
Time Frame: Up to 24 hours after the last drug administration
Population: PKA
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | PBTZ169, 160 mg | PBTZ169, 320 mg | PBTZ169, 640 mg
Number analyzed (Participants) | 4 | 4 | 5
ng*h/ml | 113.293 (73.9862) | 349.308 (282.1627) | 502.895 (167.7201)

16. Secondary Outcome: AUC (0-t)
Description: Area under the plasma concentration of PBTZ169 versus time curve in frames [0-last concentration above lower limit of quantification (LLoQ)]
Time Frame: Up to 72 hours after the last drug administration
Population: PKA
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | PBTZ169, 160 mg | PBTZ169, 320 mg | PBTZ169, 640 mg
Number analyzed (Participants) | 4 | 4 | 5
ng*h/ml | 113.259 (73.9728) | 356.170 (282.0489) | 502.075 (168.5111)

17. Secondary Outcome: AUC(0-∞) of PBTZ169
Description: Area under the plasma concentration versus time curve in frames [0-∞]
Time Frame: Up to 72 hours after the last drug administration
Population: PKA
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | PBTZ169, 160 mg | PBTZ169, 320 mg | PBTZ169, 640 mg
Number analyzed (Participants) | 4 | 4 | 5
ng*h/ml | 141.855 (87.0391) | 412.819 (299.2734) | 568.581 (189.4584)

18. Secondary Outcome: Accumulation Ratios for the PK Parameters AUC(0 -24)
Description: Accumulation ratios for the PK parameter AUC(0 -24): AUC(0- 24,ss)/AUC(0 -24), Day 1, on the original scale
Time Frame: 24 hours after the first and the last drug administration
Population: PKA
Measure: Geometric Mean (90% Confidence Interval); unit: ratio
Arm/Group | PBTZ169, 160 mg | PBTZ169, 320 mg | PBTZ169, 640 mg
Number analyzed (Participants) | 4 | 4 | 5
ratio | 1.50 [0.81 to 2.76] | 2.35 [1.28 to 4.34] | 2.74 [1.58 to 4.73]

19. Secondary Outcome: Average Concentration (Css,av) of PBTZ169
Description: Average steady-state concentration in the dosing interval following multiple dosing was evaluated as the ratio AUC0 24/τ (τ = the dosing interval)
Time Frame: Up to 72 hours after the last drug administration
Population: PKA
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | PBTZ169, 160 mg | PBTZ169, 320 mg | PBTZ169, 640 mg
Number analyzed (Participants) | 4 | 4 | 5
ng/ml | 862.63 (606.973) | 793.27 (212.270) | 532.95 (325.436)

20. Secondary Outcome: Fluctuations (%) in the Dosing Interval
Description: Fluctuations (%) in the dosing interval after multiple dosing ((Cmax - Cmin) × 100%/Css,av)
Time Frame: Up to 72 hours after the last drug administration
Population: PKA
Measure: Mean (Standard Deviation); unit: % (ratio)
Arm/Group | PBTZ169, 160 mg | PBTZ169, 320 mg | PBTZ169, 640 mg
Number analyzed (Participants) | 4 | 4 | 5
% (ratio) | 32955.25 (18636.037) | 24703.16 (19047.811) | 16253.19 (7977.030)

21. Secondary Outcome: Total (Plasma) Clearance (Clt) of PBTZ169
Description: Clt/F (apparent total clearance following single and multiple oral administration) was calculated using the following formula:
  Cl_t/F=D/AUC where D is the daily dose of the drug.
Time Frame: 24 hours after the first drug administration
Population: PKA
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | PBTZ169, 160 mg | PBTZ169, 320 mg | PBTZ169, 640 mg
Number analyzed (Participants) | 4 | 4 | 7
L/h | 3293.80 (3329.026) | 2375.06 (759.203) | 2935.49 (1382.371)

22. Secondary Outcome: Total (Plasma) Clearance (Clt) of PBTZ169
Description: as for outcome 21
Time Frame: 24 hours after the last drug administration
Population: PKA
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | PBTZ169, 160 mg | PBTZ169, 320 mg | PBTZ169, 640 mg
Number analyzed (Participants) | 4 | 4 | 5
L/h | 1393.31 (606.676) | 1200.61 (899.707) | 1259.77 (519.021)

23. Secondary Outcome: Volume of Distribution (Vd) of PBTZ169
Description: Distribution volume Vd for a dosing interval of 72 hours after the last dose
Time Frame: Up to 72 hours after the last drug administration
Population: PKA
Measure: Mean (Standard Deviation); unit: L
Arm/Group | PBTZ169, 160 mg | PBTZ169, 320 mg | PBTZ169, 640 mg
Number analyzed (Participants) | 4 | 4 | 5
L | 4.7206 (3.0828) | 14.5545 (11.7568) | 20.9540 (6.9883)

24. Secondary Outcome: Plasma Half-life Time (T1/2) of PBTZ169
Time Frame: 24 hours after the fist drug administration
Population: PKA
Measure: Mean (Standard Deviation); unit: h
Arm/Group | PBTZ169, 160 mg | PBTZ169, 320 mg | PBTZ169, 640 mg
Number analyzed (Participants) | 4 | 4 | 7
h | 10.201 (4.6319) | 16.469 (9.5669) | 10.110 (2.1530)

25. Secondary Outcome: Plasma Half-life Time (T1/2) of PBTZ169
Time Frame: 24 hours after the last drug administration
Population: PKA
Measure: Mean (Standard Deviation); unit: h
Arm/Group | PBTZ169, 160 mg | PBTZ169, 320 mg | PBTZ169, 640 mg
Number analyzed (Participants) | 4 | 4 | 5
h | 15.524 (4.0037) | 13.790 (2.3234) | 8.883 (2.5338)

26. Secondary Outcome: Elimination Constant (Kel) of PBTZ169
Description: Apparent terminal elimination rate constant was evaluated based on the regressional dependence of log-transformed concentrations ln(C) on time for the terminal log- linear part of the concentration-time curve.
Time Frame: 24 hours after the first drug administration
Population: PKA
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | PBTZ169, 160 mg | PBTZ169, 320 mg | PBTZ169, 640 mg
Number analyzed (Participants) | 4 | 4 | 7
1/h | 0.0797 (0.0371) | 0.0524 (0.0250) | 0.0708 (0.0126)

27. Secondary Outcome: Elimination Constant (Kel) of PBTZ169
Description: as for outcome 26
Time Frame: 72 hours after the last drug administration
Population: PKA
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | PBTZ169, 160 mg | PBTZ169, 320 mg | PBTZ169, 640 mg
Number analyzed (Participants) | 4 | 4 | 5
1/h | 0.0470 (0.0123) | 0.0515 (0.0098) | 0.0828 (0.0211)

ADVERSE EVENTS:
Time Frame: Collection and evaluation of safety data started at the Screening Visit (Day -10 to -1) after signing the informed consent form and was continued till the last visit of the patient within the study (Day 21+1)
Arm/Group | PBTZ169, 160 mg | PBTZ169, 320 mg | PBTZ169, 640 mg | Isoniazid, 600 mg
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/7 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 1/7 | 0/1
Other Adverse Events (participants affected / at risk) | 3/4 | 3/4 | 2/7 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PBTZ169, 160 mg (N=4) | PBTZ169, 320 mg (N=4) | PBTZ169, 640 mg (N=7) | Isoniazid, 600 mg (N=1)
Spontaneously opened tuberculous paraproctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PBTZ169, 160 mg (N=4) | PBTZ169, 320 mg (N=4) | PBTZ169, 640 mg (N=7) | Isoniazid, 600 mg (N=1)
Sinus arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Wandering atrial pacemaker (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperthermia (General disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Fever (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metabolic disorders found in ECG (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
QTc elongation (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
QTc(F) shortening (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Repolarization disturbances in the V1 lead in ECG (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Reduced (+)T amplitude in standard leads (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
ESR over 2.5 x normal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The agreements between the Principal Investigators and the CRO restricts the PIs' rights to discuss or publish trial results after the trial is completed.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-20): https://cdn.clinicaltrials.gov/large-docs/34/NCT03334734/Prot_SAP_000.pdf